CLINICAL TRIAL: NCT03924115
Title: Evaluation of a Transmedial Psychoeducational Program to Improve Pharmacological Adherence in Hypertensive Elderly Persons
Brief Title: Evaluation of a Transmedial Psychoeducational Program to Improve Pharmacological Adherence
Acronym: AFAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Concepcion (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AFAM2017; FONDEF ID16AM0007 (Other: Comisión Nacional de Ciencia y Tecnología CONICYT)
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Essential Hypertension
Keywords: Adherence, Hypertension, Mobil App, video
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Intervention Model Description: Clinical trial with a 3 parallel groups of hypertensive elderly people in 2 primary health center (CESFAM). Group A was chosen at random in CESFAM Hualpencillo, Groups B and C were selected by pairing with group A, in CESFAM Hualpencillo and Talcahuano Sur, respectively. The match was made based on 5 criteria: sex, age (± 5 years), educational level, co-morbidities (diabetes mellitus 2, chronic kidney disease and heart failure) and adherence (adherent or non-adherent). Persons who agreed to participate signed an informed consent before, to be recruited. In Group A, patients were given a smartphone with a data plan for 1 year. In each evaluations, group activities were carried out in CESFAM and home visits to those who did not attend. In each evaluation the instrument developed by the same research team was applied. For updating drugs prescription, in mobile application and collection of clinical data such as tests and controls, weekly visits were made to CESFAM.
Who Masked: Outcomes Assessor
Masking Description: Being treatment supportive care, patients and researchers know who are the participants of the different levels of intervention. The health professionals who attend both CESFAM do not have access to the information of the patients under study, as well as the evaluation of results, to avoid biases both in the care of patients and in the analysis of results. The results evaluator will receive the instrument data and validated questionnaires in previously typed code forms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Total (Experimental): This group of patients was chosen at random. They are patients who receive the full PST as intervention, that is, they receive a Smartphone with the AFAM-Health application with all the contents of the PST and data plan for 1 year.
  Interventions: Device: Transmedial Psychoeducational Program to improve adherence full or partial (PS)
- Group Partial (Experimental): This group of patients was chosen at random under the criteria of parity with group A. They are patients who receive partial PST as intervention, that is, they only receive video capsules reproduced in the CESFAM waiting room as educational content.
  Interventions: Device: Transmedial Psychoeducational Program to improve adherence full or partial (PS)
- Group Control (No Intervention): This group of patients is the control group, that is, they do not receive any type of intervention additional to the one they already receive from their CESFAM.

INTERVENTIONS:
Device: Transmedial Psychoeducational Program to improve adherence full or partial (PS) — Intervention consists of a transmedial Psychoeducational Program, which includes cognitive, behavioral and affective aspects to generate knowledge and skills that improve self-efficacy in the elderly, it is a program based on communication in health. The proposed transmedial narrative will allow older adults to assemble information from messages arranged through various media, including audiovisual capsules that will be transmitted on screens located in the Health Center and the development of a mobile application incorporated in the cellular that will be delivered with a data plan for one year. This intervention is designed to strengthen the personal resources of the elderly (such as self-efficacy, empowerment, knowledge) that promote self-care in health.
  Arms: Group Partial; Group Total

SUMMARY:
Population in Chile has experienced an accelerated process of demographic aging, which leads to changes in the composition of morbidity and mortality, with chronic noncommunicable diseases currently predominating. One of the main problems in the treatment of people with chronic and asymptomatic pathologies such as essential arterial hypertension is the lack of pharmacological adherence, where approximately 50% farewell to the treatment, while the remaining 50% partially adheres, does not adhere or interrupt within the first year.

The solution is a Psychoeducational Transmedial Program to improve pharmacological adherence (PTA), as a support to the current treatment found in centers of primary health (CESFAM).

The PTA program offers health promotion and education proposals through video capsules transmitted in CESFAM. The full PTA program also includes an AFAM-Health phone application in which older adults can know and control the administration of their medications, schedule medication registration alerts, have access to healthy life information and pathology information, Incorporated a community through a chat that generates support and accompaniment among the participants themselves.

The aim of the study is to evaluate if Transmedial Psychoeducational Program improves the pharmacological adherence of the antihypertensive treatment in elderly people receiving medical attention at CESFAM Hualpen, in Chili.

A clinical trial was conducted with 3 parallel groups of older adults diagnosed with Essential Arterial Hypertension. There were 2 treatment groups (A and B) and a control group (C). Group A was exposed to the full PTE transmedial psychoeducational program that includes a cell phone with the application developed to improve adherence and data plan. Group B received the program without the mobile application. All participants were given a Morisky-Green test to measure pharmacological adherence and an instrument developed by the clinical team to measure the biopsychosocial characteristics of elderly under study.

t is expected to find that the pharmacological adherence of those receiving the full PST is significantly superior to the control group, and those who receive the partial PST are significantly superior to the control group.

DETAILED DESCRIPTION:
The validation was carried out in two stages, before and after pilot. First, expert evaluation , in terms of five validation criteria: clarity, impartiality, relevance, and importance of each relevant question or reagents. Secondly, the results of application to pilot sample were analyzed in two ways, question by question, according to contribution of the same, and by dimensions and sub-dimensions in terms of common factors that these have.

Data collected in the instrument by interviewers is contrasted with information in the clinical file of patients. The none Data dictionary that contains detailed descriptions of each variable has been used by the registry.

Recruitment of patients: The selected patients are contacted via telephone and are summoned to a meeting at CESFAM to publicize the project, answer questions and if they wish to participate, sign informed consent. Volunteers who cannot attend these meetings are visited in their homes and the same procedure described above is performed.

Data collection: The application of the instrument is carried out by student surveyor, with home visits and paper records, trained by the research team and under the permanent supervision of 2 researchers.

Clinical data that include vital signs, exams and controls are compiled from the corresponding CESFAM, each study group having a researcher in charge. Data for medication administration are automatically registered in AFAM-Health Web App.

Data fingering: The data of the instrument recorded on paper are typed by an external professional.

Data analysis: Databases are delivered to a statistical researcher for data analysis Type of design: The comparisons to be made are of two types, between groups (Control and two treatments) and within each group (baseline measurements and measurements with intervention). In both cases, they have paired samples, since it is proposed to pair the groups.

Comparisons between groups: To calculate the sample size of each group, the specification of the correlation of scores between groups is required; but the more correlated the groups are, the smaller the sample sizes, so the worst case was chosen, that is, calculating sample sizes relative to comparison of independent samples (unpaired), a method known as "Analysis of Variance ", so that this sample is more than sufficient for any correlation achieved between groups. Under the specifications outlined above, n = 99 cases are required for each group Comparisons within the same group: To calculate the sample size of each group, it is required to specify the standard deviation of the differences, which is less than the standard deviation by itself; therefore, the same value of the standard deviation was considered, which leads to sampling sizes higher than those required, so that the calculated sample is more than sufficient for the case of interest. Under the specifications outlined above, n = 37 cases are required for each group.

In view of the above, samples of size n = 100 for each group are more than sufficient for the proposed objectives.

The statistical analysis will be developed in several stages Stage 1: Verification of the homogeneity of the groups in the pre-intervention stage, in relation to all available variables. For this purpose, it is assessed that there is, in the three groups: Equality of means of the quantitative variable Age. The statistical test is ANOVA (Alternative nonparametric Kruskal-Wallis, in the absence of normality). Equality of the proportions of the categorical variables sex, socioeconomic level, educational level, Marital status, Live children; These proportions must be similar by pairing. The statistical test is the homogeneity of Chi-Square proportions (Fisher's exact test, R-Project software).Homogeneity of variables not used in pairing. Tests analogous to those previously known (number of living children, digital literacy, etc.).

Stage 2: Once the groups are constituted according to their homogeneity with respect to the independent variables, the homogeneity of the groups in the pre-intervention stage is verified, in relation to the variables Pharmacological Adherence of the Antihypertensive Treatment (dependent) and Self-efficacy (independent ) in pre-test version. For this purpose, it will be evaluated that there is, in the three groups:

Equality of means of the quantitative variable Self-efficacy. Statistical test: ANOVA; alternative: Kruskal-Wallis.

Equality of proportions for variable Adherence. Statistical test: Square Chi; Alternative: Fisher's Exact Test.Homogeneity of the relationships between adherence and self-efficacy. Statistical test: ANOVA, two-ways (Adherence and Group). It is expected that none of the groups reflect a significant baseline relationship between these variables.

In case of lack of homogeneity, the pairing will be reviewed, to achieve homogeneous groups at the base level.

Stage 3: After 3 months of intervention (period of the first post-test measurement), the instrument is again applied to measure adherence in the three groups. At this time, the effect of desertions (dropouts) on the results of the study should be considered, verifying the homogeneity of the groups by repeating the statistical tests of stages 1 and 2 for the groups that remain in the study. If the homogeneity is altered, the complete trio linked to each subject that defects will be eliminated from the measurements. Otherwise, it continues with the groups as they are in this stage.

Stage 4: Once the groups of people who remain in the study have been defined, the effect of the intervention (in its 2 levels, A and B) must be evaluated, with respect to the results of group C (control), through measurements of the post-test third month.

For this purpose, it will be evaluated in the three groups there is:

Homogeneity of proportions for Adherence in the three groups. Statistical test: McNemar, Significant differences are expected in treatment A and eventually B, and homogeneity of the control group; Alternative: Logistic regression (covariables: Group, Basal Adherence, Baseline Self-efficacy, Response Adherence to month 3, the Group is expected to be significant).

In case of significant differences (alpha = 0.05), the effect size is evaluated, expecting greater effects in Group A, followed by B and C.

Stages 5 and 7: They coincide with stage 3, but in months 6 and 12, respectively.

Stage 6: After 6 months of intervention, defined the participants who continue in the study (by stage 5), the procedure of stage 4 is repeated, to define if there are changes in the Adherence, with respect to basal adherence and with respect to the adherence to month 3 (which is added as a covariate).

In addition, counting on Self-efficacy measurement, it is interesting to evaluate their changes:

It is verified if there is equality of means for Self-efficacy of month 6. Statistical test: ANOVA; alternative: Kruskal-Wallis. Factors: Group and Adherence to month 3, covariate: Baseline self-efficacy, with different slopes according to the group. It would be expected that there is a significant group effect and a difference in slopes.

If significant differences are found (alpha = 0.05), the groups that present these differences are evaluated. Statistical test: multiple LSD-Fisher comparisons; alternatives: non-parametric type Bonferroni (lacking normality). They also compare slopes. Statistical test: contrasts.

Step 2 is repeated for homogeneity of adherence-self-efficacy relationships. Stage 8: After 12 months of intervention, that is, at the end of the study period, stage 6 is repeated.

Stage 9: With all the data of evolution of pharmacological adherence to antihypertensive treatment by the members of the three samples and their respective self-efficacy, an analysis of repeated measures is performed. This analysis allows discriminating between individual, temporary and treatment effects; evaluating the longitudinal aspect of the intervention. It is completed by measuring again the correlation between adherence and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* People under treatment for hypertension
* Both sexes
* Older than 60 years
* Autovalent
* read and write

Exclusion Criteria:

* Under treatment for severe psychiatric pathology
* Mental retardation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Adherence | one year
  Pharmacological adherence measured with a standardized questionnaire Morisky-Green Test

SECONDARY OUTCOMES:
Disease knowledge or beliefs Disease knowledge or belief | one year
  Measured with the instrument created by study

CONTACTS AND LOCATIONS:
Overall Officials: Hans Muller, MD, Study Chair — Universidad de Concepcion
Locations (1):
- Universidad de Concepción, Concepción, Chile

IPD SHARING:
Plan to Share IPD: No